CLINICAL TRIAL: NCT05669586
Title: A Single-arm, Single-center Clinical Trial of Patient-derived Lung Cancer Organoids for Predicting Therapeutic Response in Patients With Multiline Drug-resistant Lung Cancer
Brief Title: Organoids Predict Therapeutic Response in Patients With Multi-line Drug-resistant Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Affiliated Hospital of Jiangnan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 136286
Record Dates: First submitted 2022-12-20; First posted 2023-01-03 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Lung Cancer; Organoid
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Organoid-Guided Antitumor therapy (Experimental): lung cancer specimens are obtained from lung tumor surgery or biopsy or malignant pleural effusion are used to grow organoids. Then organoids are used for drug sensitivity tests to obtain the sensitivity to drugs. Patients will receive a relatively sensitive antitumor regimen based on the test results.
  Interventions: Drug: Antitumor therapy guided by organoid drug sensitivity test
- Physician-decided Antitumor therapy (No Intervention): According to the National Comprehensive Cancer Network's (NCCN) Guidelines for lung Cancer, physicians will determine antitumor protocols or case report. They're also not sure what the drug susceptibility test says.

INTERVENTIONS:
Drug: Antitumor therapy guided by organoid drug sensitivity test — Antitumor therapy guided by organoid will be given to Multi-line Drug-resistant Non-small Cell Lung Cancer patients.
  Arms: Organoid-Guided Antitumor therapy

SUMMARY:
This is a single-center, single-arm, open and exploratory clinical study. The purpose of this study was to evaluate the consistency and accuracy of the organogenic (PDO) model for patients with lung cancer, to predict the clinical efficacy of anticancer drugs, and to speculate and select personalized treatment regiments for patients with lung cancer who are resistant to multi-line standard therapies.

DETAILED DESCRIPTION:
As for the difficult problem of drug resistance in lung cancer after multi-line therapy, there is no standard consensus in clinical diagnosis and treatment, and relevant treatment plans are still being explored and the efficacy is unknown. Patient-derived organoid cells (PDOs) have become a reliable tumor model for drugs in vitro. PDOs is a personalized tumor model with similar characteristics to the original tumor. This model can maintain the molecular and cellular composition of the original tumor, reflect the heterogeneity of the original tumor, and realize in vitro high-throughput rapid screening of drug sensitivity, accurately predict the drug response of patients, so as to provide rapid clinical drug feedback. In recent years, lung cancer organoids have also been rapidly established to reproduce the tissue structure of primary lung tumors, screen the sensitivity of therapeutic drugs, formulate lung cancer treatment programs, and realize individualized tumor treatment of lung cancer. Patients were highly matched to their PDO responses, with 84.43% accuracy, 78.01% sensitivity and 91.97% specificity.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients: ≥18 years old.
2. For non-small cell lung cancer confirmed by histology or cytology, there is no standard protocol recommendation in the guidelines for disease progression after multiline standard therapy.
3. Expected survival ≥3 months.
4. Sign informed consent.
5. The patient is willing and able to adhere to the protocol during the study, including receiving treatment and scheduled visits and examinations, including follow-up.
6. Accessible to biopsy and/or surgery sample of metastasis and/or primitive tumour
7. At least one previously unirradiated lesion that can be accurately measured at baseline with longest diameter ≥ 10 mm (must have a short lymph node excluding axis ≥ 15 mm) according to RECIST criteria with computed tomography (CT), magnetic resonance imaging (MRI) or clinical examination for accurate repeated measures. Or an unevaluable lesion, including but not limited to pleural and ascites, bone metastasis, etc.

Exclusion Criteria:

1. Participated in clinical trials of other drugs within four weeks.
2. Histologically or cytologically confirmed small cell, large cell neuroendocrine or carcinoid.
3. Not accessible to biopsy and/or surgery sample.
4. Not enough lung tissue for a histological analysis or the remaining lung tissue is not enough to perform a routine pathological analysis.
5. There are clinical symptoms or diseases of the heart that cannot be well controlled, such as: NYHA class 2 or higher heart failure, unstable angina pectoris, myocardial infarction within 1 year, clinically significant supraventricular or ventricular arrhythmia requiring treatment or intervention of patients.
6. For female subjects: should be surgically sterilized, postmenopausal patients, or agree to use a medically approved contraceptive during the study treatment period and within 6 months after the end of the study treatment period; Serum or urine pregnancy test must be negative within 7 days and must be non-nursing. Male subjects: Patients who should be surgically sterilized, or who agree to use a medically-approved contraceptive method during the study treatment period and within 6 months after the end of the study treatment period.
7. The patient has active pulmonary tuberculosis, bacterial or fungal infection (≥ grade 2 of NCI-CTC, 3rd edition); HIV infection, HBV infection, HCV infection.

   Those who have a history of psychotropic substance abuse and cannot quit or have mental disorders.
8. The subject has any active autoimmune disease or has a history of autoimmune disease (such as the following, but not limited to: interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, nephritis, hyperthyroidism, thyroid Reduced function; subjects with vitiligo or complete remission of asthma in childhood without any intervention in adulthood can be included; subjects with asthma requiring bronchodilator medical intervention are not included).
9. According to the judgment of the investigator, there are concomitant diseases that seriously endanger the patient's safety or affect the patient's completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 1 year
  Time from randomization to any disease progression and/or death, defined according to strict RECIST (Response Evaluation Criteria in Solid Tumors) v1.1. Lesion will be assessed in comparison to baseline measurements.

SECONDARY OUTCOMES:
Overall survival | 72 weeks
  Randomize time to date of death or last known alive date calculation.
Disease control rate | an average of 1 year
  The proportion of patients with a best response grade of complete response, partial response, or stable disease that has shrunk or stabilized for a period of time.
Changes in tumor volume shrinking | 6 months
  Change in tumor volume reduction from randomization to 6 months
Prediction of the response to treatment by the patient-derived organoids | 2 years
  The drug sensitivity was tested on patient-derived tumour organoids, which is compared with clinical response of the chemo- or targeted therapy treatment.
The rate of successful generation of lung cancer organoids | 2 years
  Successful generation of lung cancer organoids (growth of lung tumoral cells).

CONTACTS AND LOCATIONS:
Overall Officials: quan liu, doctor, Principal Investigator — Affiliated Hospital of Jiangnan University
Locations (1):
- Affiliated Hospital of Jiangnan University, Wuxi, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No